CLINICAL TRIAL: NCT00257751
Title: Different Regimen of Aprotinine(Trasylol) Administration in Patients Receiving
Brief Title: Different Regimen of Aprotinine(Trasylol) Administration in Patients Receiving Antiplatelet Therapy With Clopidogrel (Plavix)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Eivind Øvrum, MD, PhD, Oslo Heart Center, Rikshospitalet HF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APROT04; APROT04
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aprotinin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Aprotinine

SUMMARY:
Clopidogrel (Plavix), a platelet ADP receptor antagonist, has become the standard of care to prevent thrombosis in interventional cardiology and is increasingly being used in unstable angina and NSTEMI. An increasing number of patients are referred to emergent or urgent CABG, and several studies, as well as our own experience, have shown that preoperative administration of irreversible platelets inhibitors increase the risk of bleeding complications following CABG.

DETAILED DESCRIPTION:
Aprotinine (Trasylol) is a potent antifibrinolytic agent known to reduce bleeding after cardiac surgery. The most commeon practice is to give Trasylol in high doses immediately before surgery, during the operation, and during the first postoperative hours. However, it has also been shown that there is a hemostatic effect of the drug when given in a lower dose postoperatively, but this remains unclear.

ELIGIBILITY:
All coronary bypass operations in patients receiving Plavix within the last 7 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2004-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Perioperative bleeding
Blood transfusions
Reoperation

SECONDARY OUTCOMES:
Difference in costs related to low/high dose

CONTACTS AND LOCATIONS:
Overall Officials: Eivind Øvrum, MD, PhD, Principal Investigator — Oslo University Hospital